CLINICAL TRIAL: NCT06563271
Title: Evaluation of Analgesic Treatments for Ankle Sprains in the Emergency Department
Brief Title: Approach to Ankle Sprains in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Sarcan, Doctor, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES-Ankle
Record Dates: First submitted 2024-07-08; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Ankle Sprains
Keywords: Range of motion; Numerical Rating Scale
MeSH Terms: conditions — Ankle Injuries | interventions — dexketoprofen trometamol; Solutions; Injections; Ibuprofen; Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Dexketoprofen (Active Comparator): Dexketoprofen 50 mg will be administered parenterally (intravenously in 150 cc isotonic saline over 15 minutes infusion).
  Interventions: Drug: Dexketoprofen Trometamol 50 Mg/mL Solution for Injection; Drug: isotonic saline
- Group Ibuprofen (Active Comparator): Ibuprofen 100 mg/ml will be administered parenterally (intravenously in 150 cc isotonic saline over 15 minutes infusion).
  Interventions: Drug: Ibuprofen 100 MG/ML Solution for Injection; Drug: isotonic saline
- Group Paracetamol (Active Comparator): Paracetamol 10 mg/ml will be administered parenterally.
  Interventions: Drug: Paracetamol 10 Mg/mL Solution for Injection

INTERVENTIONS:
Drug: Dexketoprofen Trometamol 50 Mg/mL Solution for Injection — Dexketoprofen 50 mg administered parenterally (intravenously in 150 cc isotonic saline over 15 minutes infusion).
  Arms: Group Dexketoprofen
Drug: Ibuprofen 100 MG/ML Solution for Injection — Ibuprofen 100 mg/ml administered parenterally (intravenously in 150 cc isotonic saline over 15 minutes infusion).
  Group P: Paracetamol 10 mg/ml administered parenterally (intravenously in 150 cc isotonic saline over 15 minutes infusion).
  Arms: Group Ibuprofen
Drug: Paracetamol 10 Mg/mL Solution for Injection — Paracetamol 10 mg/ml administered parenterally (intravenously in 150 cc isotonic saline over 15 minutes infusion).
  Arms: Group Paracetamol
Drug: isotonic saline — Ibuprofen and dexketoprofen will be administered intravenously (IV) by mixing them into 150 cc of isotonic saline.
  Arms: Group Dexketoprofen; Group Ibuprofen

SUMMARY:
The aim of this study is to evaluate the short-term effects of routinely applied agents on pain and joint range of motion (ROM) in ankle sprains presenting to the emergency department (ED).

DETAILED DESCRIPTION:
It is aimed to examine the effects of intravenous (IV) 50 mg dexketoprofen, IV ibuprofen 400mg and IV paracetamol 10 mg on pain and joint range of motion. To determine the effects of these agents on pain, the easily applicable Numerical Rating Scale (NRS) and Wong-Baker Faces Pain Rating Scale will be used. A standard handheld half-circle goniometer will be utilized to calculate active ankle joint ROM.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older who present to the emergency department within the first 72 hours after ankle sprain.
* Grade 1 (mild) and Grade 2 (moderate) ankle sprains.
* Exclusion of fractures and dislocations (after X-ray according to Ottawa rules).
* Absence of muscle-tendon ruptures.
* Absence of vascular and nerve injuries.
* Absence of open wounds and burns.
* Stable vital signs.
* Patients who provide written and verbal consent.

Exclusion Criteria:

* Patients who did not present to the emergency department within the first 72 hours after ankle sprain.
* Grade 3 (severe) ankle sprains.
* Multiple traumas.
* Pregnancy or suspected pregnancy.
* Ankle fractures and dislocations.
* Forensic cases.
* History of previous ankle surgery or fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of multimodal treatment methods on pain in ankle sprains. | *Patient's pain level, NRS Scale: - 0 minute before treatment -15 minute after treatment -60 minute after treatment
  Numeric Rang Scale (NRS) will be used to assess effects on pain. NRS: This scale uses 11 numbers from 0 to 10 to measure pain intensity, where 0 represents "No pain" and 10 represents "Worst (unbearable) pain."
To evaluate the effectiveness of multimodal treatment methods on pain in ankle sprains. | *Wong-Baker Faces Pain Rating Scale: - 0 minute before treatment -15 minute after treatment -60 minute after treatment
  Wong-Baker FACES pain rating scale (WBS) will be used to assess effects on pain.
  WBS: This scale uses a series of faces ranging from a smiling face representing "No pain" to a crying face representing "Worst pain" to visually express the intensity of pain.
To evaluate the effectiveness of multimodal treatment methods on Range of Motion in ankle sprains. | - 0 minute ROM before treatment - 60 minute ROM after treatment
  A standard handheld goniometer will be used to calculate Range of Motion (ROM) measurements. The aim is to determine the effects of multimodal treatment methods routinely applied in emergency services on pain and range of motion and to reveal their superiority over each other, if any. (Normal ROM values: 20° for dorsiflexion, 45° for plantar flexion)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet B. Erdem, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)